CLINICAL TRIAL: NCT01883427
Title: Placebo Controlled Study Among Children Below Four Years of Age, Investigating Whether a Glucose Oxidase Nasal Spray Can Reduce Days With Upper Respiratory Tract Infection Symptoms
Brief Title: Nasal Spray With Glucose Oxidase Preventing Common Cold in Pre-school Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Krister Tano (Other)
Responsible Party: Sponsor-Investigator, Krister Tano, MD, PhD, Umeå University
Organization: Umeå University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GObarn2013
Record Dates: First submitted 2013-04-23; First posted 2013-06-21 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Upper Respiratory Tract Infections
Keywords: Days with URTI symptoms
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Glucose Oxidase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo: Saline+glucose nasal spray (Placebo Comparator): Subjects received nasal spray containing both saline+glucose twice daily for 3 months
  Interventions: Drug: Placebo
- Nasal spray with glucose oxidase+glucose (Active Comparator): Nasal spray in a bag-on-valve device with 50U/ml containing both glucose oxidase + 5% glucose in isotone saline. Dosage: One puff in each nostril twice daily for 3 months.
  Interventions: Drug: Glucose oxidase

INTERVENTIONS:
Drug: Placebo — placebo containing saline+glucose
  Other Names: Baxter Rehydrex
  Arms: Placebo: Saline+glucose nasal spray
Drug: Glucose oxidase — a hydrogen peroxide producing enzyme that creates an acidous environment to which rhinoviruses are sensitive.
  Other Names: G2133, Sigmaaldrich
  Arms: Nasal spray with glucose oxidase+glucose

SUMMARY:
To investigate if use of glucosoxidas nasal spray can reduce the number of days with upper respiratory tract infections in children beyond 4 years.

DETAILED DESCRIPTION:
Children below 4 years of age and in public day care were invited to participate in this prospective study. The children started with a visit to an ENT doctor and after inclusion the children started to spray twice daily with glucose oxidase+glucose or only saline+glucose for 3 months. During this period the parents were asked to fill in a home protocol recording upper respiratory tract symptoms as: rhinitis, cough, fever, ear ache. After 6 weeks and 12 weeks the children had scheduled visits to the ENT department, where an ENT doctor examined the throat, nasal cavity and the ear drums for otitis media. After 12 weeks of treatment a nasopharyngeal swab was taken for bacterial culture.

ELIGIBILITY:
Inclusion Criteria:

* Children below 4 years of age

Exclusion Criteria:

* None

Max Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Westman, MD, PhD, Study Chair — Västernorrlands Landsting; Marie Ryding, MD, PhD, Study Chair — Jämtlands Landsting; Anders Niklasson, MD, Study Chair — Norrbottens Landsting; Helena Toolanen, MD, Study Chair — Norrbottens Landsting
Locations (4):
- Sweden (4):
  - Öronmottagningen, Östersund
  - Öronmottagningen, Piteå
  - Öronmottagningen, Södra Sunderbyn
  - Öronmottagningen, Sundsvall

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline+Glucose Nasal Spray: Nasal spray with saline+glucose twice daily for 3 months
  Saline + glucose: A bag on valve nasal spray device containing isotone saline and 5% glucose
- Nasal Spray With Glucose Oxidase+Glucose: Nasal spray in a bag-on-valve device with 50U/ml glucose oxidase + 5% glucose in isotone saline. Dosage: One puff in each nostril twice daily for 3 months.
  Glucose oxidase: Glucose oxidase is a hydrogen peroxide producing enzyme, imitating the inhibitory effects of the normal bacterial flora of the nasopharynx
Period: Overall Study
Arm/Group | Saline+Glucose Nasal Spray | Nasal Spray With Glucose Oxidase+Glucose
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pre-school children
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline+Glucose Nasal Spray | Nasal Spray With Glucose Oxidase+Glucose | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: months] | 28 [14 to 43] | 27 [11 to 44] | 28 [11 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  Sweden | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Infectious Symptoms
Description: Days with upper respiratory tract infection symptoms during a 3 months period are recorded in a home protocol by the parents of the children.
Time Frame: 3 months of recording
Population: Only a total of 40 Children fulfilled the study, which means that the Power are to low.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Saline+Glucose Nasal Spray | Nasal Spray With Glucose Oxidase+Glucose
Number analyzed (Participants) | 20 | 20
days
  Days with URTI | 9 (4) | 13 (10)
  Days with rhinitis | 10 (6) | 13 (10)
  Days with cough and rhinitis | 6 (5) | 8 (6)
  days with fever | 3 (3) | 5 (4)
Statistical Analysis 1: Comparison: Saline+Glucose Nasal Spray vs Nasal Spray With Glucose Oxidase+Glucose; Too few included to reach power; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — Not significant

ADVERSE EVENTS:
Time Frame: During the study period of 3 months
Arm/Group | Saline+Glucose Nasal Spray | Nasal Spray With Glucose Oxidase+Glucose
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saline+Glucose Nasal Spray (N=20) | Nasal Spray With Glucose Oxidase+Glucose (N=20)
local side effects (Respiratory, thoracic and mediastinal disorders) | 0 | 0 — Local side effects in the nasal cavity

LIMITATIONS AND CAVEATS:
We wanted 200 Children but only 40 fulfilled the study, which make the results hard to evaluate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No